CLINICAL TRIAL: NCT00513773
Title: Inflammation and Risk Prediction in Patients With Abdominal Aortic Aneurysm
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 070535; LCIC Future Leaders in CV
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Abdominal Aortic Aneurysm,; Inflammation and Risk Prediction; Diagnostic Tool Efficacy
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum/plasma for biomarker analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand the role of inflammation in the pathophysiology of abdominal aortic aneurysm. In this study we hope to show better ways of predicting risk in this condition by using a combination of FDG-PET with CT.

DETAILED DESCRIPTION:
Cumulative experimental and pathological evidence support the postulate that inflammation may serve as the unifying concept in the pathogenesis of atherosclerosis and its complications. Aneurysmal disease is associated with inflammatory cell infiltrate and enzymatic degradation of the vessel wall. Although the risk of abdominal aortic aneurysm (AAA) rupture relates to the maximum cross-sectional diameter, rapid expansion of the aortic diameters preceding fissuration and rupture has been observed in AAA independently of their initial size. However, current diagnostic modalities stratify risk of AAA rupture based solely on the size of the aneurysm without factoring potentially useful information derivable from the degree of aneurysmal wall inflammatory response.

We propose to utilize fluorodeoxyglucose (FDG) positron emission tomography (PET) imaging co-registered with structural computerized tomography (CT) images for the in vivo localization and quantification of vascular inflammation in patients with AAA in order to determine whether increased inflammation within the walls of the aneurysm correlates with rapid enlargement of AAA (change in aneurysmal diameter within 6 months), symptoms, thrombosis, or intervention for ruptured, leaking, rapidly expanding, or painful AAAs.

In patients with underlying abdominal aortic aneurysm (AAA), the progression of disease i.e. expansion is associated with increased inflammation within the aneurysm wall as characterized by FDG-PET/CT, and the degree of inflammation is a risk predictor for adverse events.

Prior studies have demonstrated that FDG uptake is greater in inflamed tissues, such as infectious foci and tumors. In chronic inflammatory lesions and malignancies, FDG uptake is increased in macrophage-dense regions. The relatively high uptake of FDG by macrophages is attributed to the relatively high metabolic rates of macrophages, and the inability of macrophages to store glycogen, making them more reliant upon external glucose as a source of fuel. Activation of macrophages can further increase their glucose consumption. Both in animal models and humans, inflamed blood vessels have been shown to have an increased uptake of FDG. Several investigators have shown that FDG-PET can reliably detect inflammation in atherosclerosis. Thus detection of enhanced FDG uptake in the aneurysmal walls of patients with AAA may have potential significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AAA between 3 to 5 cm
* Patients with AAA > 5cm in whom the risk of operative intervention is prohibitive in the opinion of the surgeon.
* No allergies to iodinated contrast.
* Diabetic patients will be eligible for this study. Patient on metformin will be asked not to take the drug for one day prior to and for two days after the procedure.
* Subjects must be able to give informed consent

Exclusion Criteria:

* Patients with an impaired kidney function, significantly elevated creatinine levels after angiography/PCI (serum creatinine level >1.5 mg/dl) will be excluded form the study.
* Unstable patients or those with decompensated heart failure will be excluded because of safety reasons.
* Pregnant or lactating women will be excluded. Pregnancy will need to be tested in all pre-menopausal women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Give more details that may enable us to better assess the chance of AAA expansion or rupture | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Uchechukwu Sampson, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States